CLINICAL TRIAL: NCT01890694
Title: Tolvaptan to Reduce Length of Stay in Hospitalized Patients With Cirrhosis and Hyponatremia
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Otsuka America Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10-02496
Record Dates: First submitted 2012-06-20; First posted 2013-07-02 (Estimated); Results first posted 2016-04-11 (Estimated); Last update posted 2017-12-11 (Actual); Status verified 2017-11

CONDITIONS: Hyponatremia
Keywords: Hyponatremia; Dilutional Hyponatremia; Euvolemic Hyponatremia; Hypervolemic Hyponatremia; Fluid Restriction; Tolvaptan
MeSH Terms: conditions — Hyponatremia | interventions — Tolvaptan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Subjects will receive placebo once daily.
  They will undergo the following procedures in every visit: Vitals (blood pressure, heart rate, respiration, temperature, weight, height), Laboratory Tests (chemistry, hematology, liver function, urine electrolytes, renin, and copeptin), ascites assessment, evaluation for edema. Quality of life assessments (SF-36, and LDQOL 1.0) will be administered on Day 1, Discharge day, Weeks 1-4 post-discharge, and months 2-6 post-discharge. Hepatic encephalopathy assessment (Number Connection Test, Digit symbol test, Constructional apraxia, Inhibitory control test, Repeatable Battery for the Assessment of Neuropsychological Status) will be administered on Days 1, 2, 4, 6, and 8; discharge day; Weeks 1-4 post-discharge; and Months 2-6 post-discharge.
  Interventions: Drug: Placebo; Behavioral: Hepatic Encephalopathy Assessment; Behavioral: Quality of Life Assessment; Biological: Vital signs; Biological: Blood laboratory tests; Procedure: Ascites Evaluation; Procedure: Edema
- Tolvaptan (Experimental): Subjects will receive Tolvaptan once daily.
  They will undergo the following procedures in every visit: Vitals (blood pressure, heart rate, respiration, temperature, weight, height), Laboratory Tests (chemistry, hematology, liver function, urine electrolytes, renin, and copeptin), ascites assessment, evaluation for edema. Quality of life assessments (SF-36, and LDQOL 1.0) will be administered on Day 1, Discharge day, Weeks 1-4 post-discharge, and months 2-6 post-discharge. Hepatic encephalopathy assessment (Number Connection Test, Digit symbol test, Constructional apraxia, Inhibitory control test, Repeatable Battery for the Assessment of Neuropsychological Status) will be administered on Days 1, 2, 4, 6, and 8; discharge day; Weeks 1-4 post-discharge; and Months 2-6 post-discharge.
  Interventions: Drug: Tolvaptan; Behavioral: Hepatic Encephalopathy Assessment; Behavioral: Quality of Life Assessment; Biological: Vital signs; Biological: Blood laboratory tests; Procedure: Ascites Evaluation; Procedure: Edema

INTERVENTIONS:
Drug: Tolvaptan — 15 mg once daily
  Arms: Tolvaptan
Drug: Placebo — 15 mg once daily
  Arms: Placebo
Behavioral: Hepatic Encephalopathy Assessment — The Number connection test, Digit symbol test, Constructional apraxia, Inhibitory control test, Repeatable Battery for the Assessment of Neuropsychological Status will be administered on Days 1, 2, 4, 6, and 8; discharge day; Weeks 1-4 post-discharge; and Months 2-6 post-discharge.
Behavioral: Quality of Life Assessment — The SF-36 and Liver Disease Questionnaire will be administered on Day 1, Discharge day, Weeks 1-4 post-discharge, and months 2-6 post-discharge
Biological: Vital signs — Vital signs (blood pressure, heart rate, respiration, temperature, weight, height) will be recorded at every visit.
Biological: Blood laboratory tests — Blood laboratory tests (chemistry, hematology, liver function, urine electrolytes, renin, and copeptin) will be recorded at every visit.
Procedure: Ascites Evaluation — Ascites will be assessed at every visit.
Procedure: Edema — Edema will be assessed at every visit.

SUMMARY:
Hyponatremia is a condition in which there is a low sodium level in the blood. Individuals with cirrhosis may develop low blood sodium as a complication of their liver disease. In these patients, the presence of low blood sodium may exacerbate other complications such as encephalopathy, resulting in confusion, drowsiness, or coma. It may also affect the ability of the body to fight infection. In certain cases, cirrhotic patients may be hospitalized for the treatment of their low blood sodium.

The drug tolvaptan is currently FDA approved for the treatment of hyponatremia in patients with cirrhosis. Although it has been shown to increase the sodium level, the clinical trials that led to its approval did not otherwise assess clinical benefit of the drug.

This study is designed to determine whether patients with cirrhosis derive a clinical benefit when they receive tolvaptan for the treatment of hyponatremia within 2 days of admission. Specifically, whether it is associated with shortened length of stay and improvement in other complications of cirrhosis.

DETAILED DESCRIPTION:
As per hyponatremia standard treatment of care, all patients considered for the study will have had diuretic therapy discontinued for at least 1 day prior to the screening visit and received volume expansion with 25% salt poor albumin, if clinically indicated to ensure adequate intravascular volume expansion as standard of care for a patient hospitalized for complications of cirrhosis.

Patients will be approached and presented with a written consent form during the first 24 hours of their admission to NYUMC (Tisch Hospital). They will be verbally informed about the purpose and procedures of the study, as well as its potential risks and benefits. Following written consent, the patients will undergo a series of screening procedures, including physical examination, medical history, blood work, and hepatic encephalopathy assessment, to determine their eligibility.

After screening and determination that the patient fulfills all inclusion and exclusion criteria, the patients will be randomized the following day on Day 0 to receive oral tolvaptan or placebo once daily. Patients in the treatment arm will receive oral tolvaptan at an initial dose of 15mg once daily. The placebo arm will be used as a comparison group to determine whether long-term, ambulatory tolvaptan administration is associated with clinical benefits to patients with cirrhosis and hyponatremia. Patients in the placebo arm will receive current standard of treatment for patients with cirrhosis and hyponatremia. Current standard treatment of hyponatremia in cirrhotic patients involves fluid restriction in the diet (1L fluid daily), discontinuation of diuretic therapy (such as furosemide, spironolactone), and frequent monitoring of the sodium level. Severe hyponatremia (Na<120mEq/L) involves infusion of hypertonic saline.

Patients will be encouraged to drink in response to thirst, and patients will be re-evaluated at 8 hours with determination of Na level after the first dose. If the serum sodium concentration remains below 136 mEq/L or increases by less than 5 mEq/L during the prior 24 hours, the dose will be increased from 15mg to a maximum dose of 30mg. Too rapid correction of serum sodium will be defined as either 8 mEq/L in the first 8 hours or greater than 12mEq/L over 24 hours. In these situations, tolvaptan will either be withheld or decreased at the next dose or the patient instructed to increase fluid intake. Similar adjustments will be made if the serum sodium concentration rises above 145mEq/L.

Patients will undergo a physical examination and laboratory evaluation that will include electrolytes, BUN/Cr, and liver tests and determination for reason for continued hospitalization as per standard of care from Day 1 to 8 or until day of discharge if discharge occurs prior to Day 8. Neutrophil function assay will be obtained upon randomization and at week 4 after discharge. Urine electrolytes and renin and copeptin levels will be obtained at Day 0, Day 8 (if still hospitalized), day of discharge, and monthly.

Patients will undergo a detailed assessment for hepatic encephalopathy on Days 0, 2, 4, and 8 or until day of discharge if it occurs prior to Day 8. Patients will also have a complete assessment on day of discharge if occurs after Day 8. Quality of life questionnaires will be completed at Day 0, Day 8 (optional), day of discharge (optional), and weekly for the first month and then monthly for a total of 3 months after discharge. In addition, patients will be asked to complete the questionnaires during their follow-up visits, which will occur 1, 2, and 4 weeks after study drug discontinuation.

Patients with clinically significant fluid overload (moderate ascites, grade 1 edema), Na level 130 or greater, asterixis is not present, and severe azotemia is not present (BUN less than 30mg/dl, Cr less than 1.5mg/dl) will be started on spironolactone 50mg daily and furosemide 20mg daily. Doses will be increased by 50mg and 20mg, respectively, daily every week if clinically significant fluid overload persists, weight loss over the previous week was less than 5 lbs, and the above safety assessments remain satisfied. Diuretic doses will be either reduced or held for excessive fluid loss (more than 10 lbs over the previous week) or one of the safety parameters are present.

At discharge, patients will continue on Study Drug with weekly visits for one month and then monthly, after discharge, for 3 months. At each visit, patients will have an interim history (need for hospitalization), performance of large volume paracentesis and volume of ascites removed, physical examination, liver and kidney tests, and assessment of hepatic encephalopathy.

Following the discontinuation of the study drug, patients will be asked to come to the clinic for follow-up visits at weeks 1, 2, and 4, post-discontinuation of study drug. At each visit, patients will have an interim history (need for hospitalization), performance of large volume paracentesis and volume of ascites removed, physical examination, liver and kidney tests, and assessment of hepatic encephalopathy.

ELIGIBILITY:
Inclusion Criteria:

* Cirrhosis
* Screening within 24 hours of admission
* Na level less than 130mEq/L
* Presence of fluid overload with either history of ascites or edema
* Cr < 2.0mg/dl
* Planned length of stay after randomization of at least 24 hours
* Anticipated survival of at least 8 days
* Ability to provide informed consent

Exclusion Criteria:

* Hospitalization greater than 24 hours at screening
* Depletional hyponatremia
* Hyponatremia due to hyperglycemia
* Acute and transient hyponatremia associated with head trauma or post-operative states
* Hyponatremia due to primary polydipsia, adrenal insufficiency, or hypothyroidism
* Urgent need for treatment of hyponatremia with saline or hypertonic saline
* Treatment with demeclocycline, lithium chloride, and urea
* Cr greater than 2.0mg/dl
* Stage 3 or 4 hepatic encephalopathy
* Inability to provide informed consent
* Planned discharge within 24 hours
* Anticipated survival less than 8 days
* GI bleeding within one month of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2012-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Sigal, MD, Principal Investigator — NYU School of Medicine
Locations (1):
- NYU Langone Medical Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Subjects will receive placebo once daily.
- Tolvaptan: Subjects will receive 15 mg Tolvaptan once daily.
Period: Overall Study
Arm/Group | Placebo | Tolvaptan
Started | 1 | 1
Completed | 0 | 0
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Tolvaptan | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Length of Hospital Stay
Description: Performance period for sponsored trial expired and not enough subjects were enrolled in study. Funding sponsor did not continue support.
Time Frame: participants will be followed for the duration of hospital stay, an expected average of 2 weeks
Population: Data were not collected due to premature termination of the trial
Arm/Group | Placebo | Tolvaptan
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Severity of Hepatic Encephalopathy
Description: Change from baseline of Hepatic Encephalopathy
Time Frame: Day 2
Population: Performance period for sponsored trial expired and not enough subjects were enrolled in study. Funding sponsor did not continue support.
Groups:
- Tolvaptan: Subjects will receive Tolvaptan once daily.
- Placebo: Study Terminated. No data analyzed
Arm/Group | Tolvaptan | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Severity of Hepatic Encephalopathy
Description: Change from baseline of Hepatic Encephalopathy
Time Frame: Day 4
Population: as for outcome 2
Arm/Group | Tolvaptan | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Severity of Hepatic Encephalopathy
Description: Change from baseline of Hepatic Encephalopathy
Time Frame: Day 6
Population: as for outcome 2
Arm/Group | Tolvaptan | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Severity of Hepatic Encephalopathy
Description: Change from baseline of Hepatic Encephalopathy
Time Frame: Day 8
Population: as for outcome 2
Arm/Group | Tolvaptan | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Severity of Hepatic Encephalopathy
Description: Change from baseline of Hepatic Encephalopathy
Time Frame: participants will be followed for the duration of hospital stay, an expected average of 2 weeks
Population: as for outcome 2
Arm/Group | Tolvaptan | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Severity of Hepatic Encephalopathy
Description: Change from baseline of Hepatic Encephalopathy
Time Frame: Week 1-4 Post-discharge
Population: as for outcome 2
Arm/Group | Tolvaptan | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Severity of Hepatic Encephalopathy
Description: Change from baseline of Hepatic Encephalopathy
Time Frame: Months 2-6 post-discharge
Population: as for outcome 2
Arm/Group | Tolvaptan | Placebo
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Ascites
Description: Improved control of ascites
Time Frame: Day 1 to Post-discharge (6 months)
Population: as for outcome 2
Arm/Group | Tolvaptan | Placebo
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Renal Function [BUN and Creatinine Laboratory Results]
Description: Improved renal function from baseline
Time Frame: Day 1 to Post-discharge (6 months)
Population: as for outcome 2
Arm/Group | Tolvaptan | Placebo
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Hospital Readmission Rate
Description: Lower readmission rate
Time Frame: Post-Discharge (6 months)
Population: as for outcome 2
Arm/Group | Tolvaptan | Placebo
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Survival
Description: Improved chances of survival when receiving Tolvaptan vs. standard of care
Time Frame: Post-discharge (6 months)
Population: as for outcome 2
Arm/Group | Tolvaptan | Placebo
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Neutrophil Function [Results From the Assay of Neutrophils]
Description: Improved neutrophil function from baseline
Time Frame: Day 1 to Post-discharge (6 months)
Population: as for outcome 2
Arm/Group | Tolvaptan | Placebo
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Tolerability of Diuretic Therapy
Description: Improved ability to tolerate diuretic therapy, as evidenced by reduced adverse events to diuretic therapy and reduced risk of re-hospitalization.
Time Frame: Day 1 until Discharge (participants will be followed for the duration of hospital stay, an expected average of 2 weeks)
Population: as for outcome 2
Arm/Group | Tolvaptan | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Placebo | Tolvaptan
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1

LIMITATIONS AND CAVEATS:
Due to the small sample size, data was not able to be analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No